CLINICAL TRIAL: NCT01179919
Title: Oseltamivir and Oseltamivir Carboxylate Pharmacokinetics in Obese Adults
Brief Title: Pharmacokinetics of Oseltamivir Carboxylate In Morbidly Obese Subjects
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Manjunath Prakash Pai (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor-Investigator, Manjunath Prakash Pai, Associate Professor, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 10-002
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Results first posted 2016-12-06 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Obesity
Keywords: Oseltamivir; Obesity; Influenza; Pharmacokinetics in Obesity
MeSH Terms: conditions — Obesity; Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oseltamivir Dosed Group (Experimental): Oseltamivir 75 mg by mouth every 12 hours for 9 doses
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Oseltamivir — Capsule, 75 mg by mouth for 9 doses
  Other Names: Tamiflu

SUMMARY:
One in three Americans are obese. Obese subjects may or may not need higher doses of the anti-flu drug known as Tamiflu (oseltamivir). The current study is being done to see if the FDA approved dose of oseltamivir will achieve similar concentrations in obese healthy volunteers compared to that previously shown in non-obese volunteers.

DETAILED DESCRIPTION:
The incidence of obesity has increased dramatically over the past two decades in the United States (US). Twenty-five percent of adult Americans are now classified as obese. Obesity is associated with physiological alterations that can affect drug clearance and volume of distribution. Obese subjects are often excluded from phase 1 pharmacokinetic studies. As a result, drug dosing regimens developed for clinical use may not be appropriate for the obese population. Use of fixed dosing regimens may result in under dosing of obese patients. In contrast adjustment of drug dosing based on total body weight may lead to over dosing of obese patients. Oseltamivir phosphate (Tamiflu®) is an antiviral agent that is currently dosed as 75 mg once daily for chemoprophylaxis and twice daily for treatment of influenza in adults.

Oseltamivir is rapidly converted to its active metabolite, oseltamivir carboxylate by esterases. The clearance of oseltamivir carboxylate is dependent on tubular secretion and glomerular filtration. Given that these drug elimination pathways may be enhanced in obese individuals, oseltamivir carboxylate plasma exposures may be lower in obese subjects compared to normal weight subjects. Although a specific plasma exposure target for oseltamivir carboxylate has not been established, lower oseltamivir carboxylate exposures may predispose obese patients to treatment failure and increase the probability for emergence of oseltamivir-resistant influenza virus. The current study proposes to characterize the plasma oseltamivir carboxylate concentration-time profile after multiple doses of oral oseltamivir in a cohort of healthy morbidly obese subjects. The study will be performed using a phase 1, open-label,multiple dose, pharmacokinetic study design in twenty obese adult subjects. This pilot study will provide pharmacokinetic data that may be incorporated into existing oseltamivir carboxylate population pharmacokinetic models to define appropriate doses of oseltamivir in obese patients.

ELIGIBILITY:
Inclusion Criteria:

* males and females, 18 to 50 years of age
* non-smoking or light-smoking (≤5 cigarettes per day) volunteers
* BMI ≥ 40 kg/m2
* female subjects of childbearing potential either surgically sterilized, using an effective method of contraception (diaphragm, cervical cap,condom) or agree to abstain from sex from time of pre-study screening, during entire study period and 1 week following the study period.

Exclusion Criteria:

* history of significant hypersensitivity reaction to oseltamivir
* history of gastric bypass surgical procedure
* history of significant clinical illness requiring pharmacological management
* abnormal serum electrolyte or complete blood count requiring further clinical work-up
* transaminases (AST or ALT) >2.5 x upper limit of normal
* estimated creatinine clearance <50 mL/min (Cockcroft-Gault equation)
* positive urine pregnancy test (if female)
* abnormal electrocardiogram (ECG) as judged by study physician
* unable to tolerate venipuncture and multiple blood draws
* clinically significant abnormal physical examination defined as a physical finding requiring further clinical work-up

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2010-07; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manjunath Pai, PharmD, Principal Investigator — ACPHS
Locations (1):
- TKL Research, Paramaus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
The summative data have been published and are available as open-access to the public: doi10.1128/AAC.00422-11

REFERENCES:
- [Derived] Pai MP, Lodise TP Jr. Oseltamivir and oseltamivir carboxylate pharmacokinetics in obese adults: dose modification for weight is not necessary. Antimicrob Agents Chemother. 2011 Dec;55(12):5640-5. doi: 10.1128/AAC.00422-11. Epub 2011 Sep 19. PMID 21930881

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oseltamivir Dosed Group
Started | 21
Completed | 19
Not Completed | 2
Not completed — Protocol Violation | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Subjects administered at least 1 dose of oseltamivir
Arm/Group | Oseltamivir Dosed Group
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 36 [19 to 50]
Gender [Count of Participants; unit: Participants]
  Female | 17
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 11
  More than one race | 3
  Unknown or Not Reported | 0
Body Mass Index [Median (Full Range); unit: kg/m^2] | 43.7 [40.0 to 54.4]

OUTCOME MEASURES:

1. Primary Outcome: Steady-State AUC of Oseltamivir Carboxylate
Description: AUC is the area under the concentration-time curve. This is measured as concentration in nanograms of oseltamivir carboxylate per milliliter of plasma multiplied by time in hours (hour*ng/mL)
Time Frame: 6 days
Population: Subjects who received all 9 doses of oseltamivir
Measure: Mean (Standard Deviation); unit: hour*ng/mL
Arm/Group | Oseltamivir Dosed Group
Number analyzed (Participants) | 19
hour*ng/mL | 2579 (510)

2. Secondary Outcome: Steady-State Cmax and Cmin of Oseltamivir Carboxylate
Description: Cmax is the maximum concentration and Cmin in the minimum concentration of oseltamivir carboxylate measured in nanogram of oseltamivir carboxylate per milliliter of plasma (ng/mL)
Time Frame: 6 days
Population: Subjects who received all 9 doses of oseltamivir
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Oseltamivir Dosed Group
Number analyzed (Participants) | 19
ng/mL
  Cmax | 316 (68.1)
  Cmin | 113 (37.4)

ADVERSE EVENTS:
Time Frame: 6 days
Arm/Group | Oseltamivir Dosed Group
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oseltamivir Dosed Group (N=21)
Anxiety (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study only evaluated obese subjects. The concentrations measured in plasma may not reflect concentrations in tissues such as the lungs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No